CLINICAL TRIAL: NCT02645214
Title: Antiseptic Scrub Contamination and Transmission Trial: A Randomized Controlled Trial to Evaluate the Impact of Antiseptic Scrubs on Bacterial Contamination.
Brief Title: Antiseptic Scrub Contamination and Transmission Trial
Acronym: ASCOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00062781
Record Dates: First submitted 2015-12-31; First posted 2016-01-01 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2016-03

CONDITIONS: Disease Transmission

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control scrubs (non-antiseptic) (Placebo Comparator): subject will wear control scrubs for the duration of a 12-hour ICU shift
  Interventions: Other: Non-antiseptic scrubs
- Antiseptic Impregnated Scrubs Type 1 (Active Comparator): subject will wear antiseptic impregnated scrubs-type 1 for the duration of a 12-hour ICU shift
  Interventions: Other: Antiseptic scrubs
- Antiseptic Impregnated Scrubs Type 2 (Active Comparator): subject will wear antiseptic impregnated scrubs-type 2 for the duration of a 12-hour ICU shift
  Interventions: Other: Antiseptic scrubs

INTERVENTIONS:
Other: Non-antiseptic scrubs
  Arms: Control scrubs (non-antiseptic)
Other: Antiseptic scrubs
  Arms: Antiseptic Impregnated Scrubs Type 1; Antiseptic Impregnated Scrubs Type 2

SUMMARY:
This study is a prospective, blinded, randomized, controlled trial (RCT) with a crossover design to determine if antiseptic-impregnated surgical scrubs decrease the burden of healthcare providers (HCP) clothing contamination compared to standard, control surgical scrubs following a 12-hour ICU shift.

DETAILED DESCRIPTION:
The investigators will perform a 3-arm prospective, blinded, randomized, controlled trial with a cross-over design to determine if HCP who wear antiseptic-impregnated clothing (i.e., surgical scrubs) will acquire and transmit fewer pathogens than HCP wearing standard clothing.

A total of 40 intensive care unit (ICU) nurses (from the Medical and Surgical ICUs in the Duke Medical Pavilion) will be enrolled and sign a consent form to participate in the study. Their main task will be to wear control (non- antiseptic) scrubs (Arm 1) and two different types of antiseptic-impregnated scrubs (Arms 2 and 3). Subjects will be randomized to one of 6 strategies. Each nurse typically cares for two patients each day and will be enrolled for three consecutive days (or shifts, if they do not work for 3 days in a row). Once the nurses have consented to participate in this project, the study coordinator will provide the 3 sets of scrubs and will label them with numbers, thus blinding the nurses to which scrubs they will wear on which day. The nurse will wear the scrubs on the 3 pre-arranged shifts.

Data will be summarized using standard statistical methods. The investigators will utilize linear mixed models to compare relative differences in the amount of contamination between arms at the end of the shift to adjust for our crossover study design. Mixed effects logistic regression models will be used to compare proportions. All calculations will be adjusted for the amount of environmental contamination observed during the shift and contamination on HCP clothing in the beginning of the shift. Statistical significance for two primary comparisons (each antiseptic scrub versus control) will be corrected for multiple comparisons.

This is a minimal risk study and the investigators have no safety concerns from the patients or nurses as relates to obtaining swabs and room cultures, nor with wearing the scrubs and having them cultured. Data will be stored on encrypted Duke Medicine servers (participant log & study IDs) and/or in our REDCap database (all other data collected for the study).

ELIGIBILITY:
Inclusion Criteria:

* All intensive care unit (ICU) nurses at Duke Medical Center are eligible to participate in this study.

Exclusion Criteria:

* Nurses outside the Duke Medical Center ICU will not be eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
The difference in total acquired contamination (Total CFU) on HCP clothing at the end of a 12-hour ICU shift. | At the end of a 12-hour ICU shift

SECONDARY OUTCOMES:
The presence or absence of individual specific pathogens: S. aureus (MRSA or MSSA), Enterococci (VRE or VSE), Acinetobacter spp., Pseudomonas spp., and Enterobacteriaceae of interest such as E. coli and Klebsiella spp. | At the end of a 12-hour ICU shift
The proportion of positive cultures - overall and at each culture location | At the end of three 12-hour ICU shifts
The number of suspected and confirmed "transmission events" | At the end of three 12-hour ICU shifts
The proportion of suspected and confirmed "transmission events" | At the end of three 12-hour ICU shifts
Health care personnel perceptions of clothing as measured by survey | At the end of a 12-hour ICU shift

CONTACTS AND LOCATIONS:
Overall Officials: Deverick Anderson, MD, MPH, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Derived] Anderson DJ, Addison R, Lokhnygina Y, Warren B, Sharma-Kuinkel B, Rojas LJ, Rudin SD, Lewis SS, Moehring RW, Weber DJ, Rutala WA, Bonomo RA, Fowler VG, Sexton DJ; CDC Prevention Epicenters Program. The Antimicrobial Scrub Contamination and Transmission (ASCOT) Trial: A Three-Arm, Blinded, Randomized Controlled Trial With Crossover Design to Determine the Efficacy of Antimicrobial-Impregnated Scrubs in Preventing Healthcare Provider Contamination. Infect Control Hosp Epidemiol. 2017 Oct;38(10):1147-1154. doi: 10.1017/ice.2017.181. Epub 2017 Aug 29. PMID 28847326